CLINICAL TRIAL: NCT00109122
Title: A Double-Blind, Placebo-Controled, Randomized Study to Evaluate Safety, Tolerability, and Immunogenicity After 1 and 2 Doses of Zoster Vaccine
Brief Title: Safety, Tolerability, and the Body's Ability to Develop Resistance to an Investigational Vaccine for Shingles (V211-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-007; 2005_017
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Biological: zoster vaccine live (Oka/Merck)
  Other Names: V211
Biological: Comparator: placebo (unspecified)

SUMMARY:
The purpose of this study is to determine the immunity (the body's protection) against shingles after receiving two doses of an investigational vaccine or placebo (a look alike vaccine with no active ingredients).

DETAILED DESCRIPTION:
The duration of treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are at least 60 years of age with a history of varicella (shingles)
* Females must have been postmenopausal.

Exclusion Criteria:

* Subjects who did not previously participate in the main study of this protocol.
* Subject had shingles since their 6 month follow-up visit in main phase of study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2001-11; Primary Completion 2003-02 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
VZV ELISPOT response ~6 weeks after 1 and 2 doses | 6 weeks after 1 and 2 doses

SECONDARY OUTCOMES:
To assess the safety and tolerability of the zoster vaccine. To evaluate the long-term persistence of the VZV-specific cell mediate immunity and the VZV-specific antibody response at 1 through 3 years after 2 doses of vaccine or placebo | 1 through 3 years after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Vermeulen JN, Lange JM, Tyring SK, Peters PH, Nunez M, Poland G, Levin MJ, Freeman C, Chalikonda I, Li J, Smith JG, Caulfield MJ, Stek JE, Chan IS, Vessey R, Schodel FP, Annunziato PW, Schlienger K, Silber JL. Safety, tolerability, and immunogenicity after 1 and 2 doses of zoster vaccine in healthy adults >/=60 years of age. Vaccine. 2012 Jan 20;30(5):904-10. doi: 10.1016/j.vaccine.2011.11.096. Epub 2011 Dec 7. PMID 22154769
- Available data/document: CSR Synopsiis — http://www.merck.com/clinical-trials/policies-perspectives.html